CLINICAL TRIAL: NCT01853150
Title: Repetitive Transcranial Magnetic Stimulation for Freezing of Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dongtan Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Suk Yun Kang, MD, PhD, Dongtan Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-022
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Parkinsonian Disorders
MeSH Terms: conditions — Parkinsonian Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS Motor cortex (Experimental): rTMS will be applied over the motor cortex
  Interventions: Device: rTMS Motor cortex
- rTMS Supplementary motor area (Active Comparator): rTMS will be applied over the supplementary motor area
  Interventions: Device: rTMS Supplementary motor area

INTERVENTIONS:
Device: rTMS Motor cortex
  Arms: rTMS Motor cortex
Device: rTMS Supplementary motor area
  Arms: rTMS Supplementary motor area

SUMMARY:
Freezing of gait (FOG) means that patients cannot walk without any known causes, other than parkinsonism, which is very disabling symptom. Patients descirbe their feeling of the feet suddenly being glued to the floor. Transcranial magnetic stiumation is a noninvasive procedure using electromagnetic induction to stimulate brain. Transcranial magnetic stiumation (rTMS) can selectively change brain activity to enhance desired effects. The aim of this study is to the therapeutic effect of rTMS for the FOG.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease or Primary progressive freezing of gait
* age 18 and older
* Freezing of gait

Exclusion Criteria:

* pregnant or any, other medical, surgical, neurological or psychiatric conditions
* other restrictions which prevent you from undergoing TMS recording, such as; surgically or traumatically implanted foreign bodies such as a pacemaker, an implanted medication pump, a metal plate in the skull, or metal inside the skull or eyes (other than dental appliances or fillings), and/ or heart/cardiac lines
* any past or current history of seizure disorder or epilepsy
* unable to give informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
The number of steps | 2 days
  The number of steps during the stand-walk-sit (SWS) test

SECONDARY OUTCOMES:
The completion time during the SWS test | 2 days
Freezing episodes of gait trajectory | 2 days
Patient and Clinical Global Impression Scale | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do, South Korea